CLINICAL TRIAL: NCT05198791
Title: The Effect of Mineralocorticoid Receptor Antagonist Therapy in Patients with Acute Myocardial Infection or Injury and Cardiovascular Risk Factors: a Registry-based, Stratified-medicine, Randomised, Controlled Trial
Brief Title: Stratified Medicine of Eplerenone in Acute MI/injury (StratMed-MINOCA)
Acronym: StratMedMINOCA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NHS National Waiting Times Centre Board (Other)
Collaborators: British Heart Foundation (Other); Abbott (Industry)
Responsible Party: Principal Investigator, Colin Berry, Professor, NHS National Waiting Times Centre Board
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: StratMed-MINOCA
Record Dates: First submitted 2021-12-20; First posted 2022-01-20 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Myocardial Infarction, Acute; Myocardial Infarction with Nonobstructive Coronary Arteries; Myocardial Injury
Keywords: Stratified Medicine; Mineralocorticoid receptor antagonists; MINOCA; Myocardial injury; Myocardial infarction; Myocardial Infarction with Nonobstructive Coronary Arteries
MeSH Terms: conditions — Myocardial Infarction; MINOCA | interventions — Tablets; Eplerenone; Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, open-label, blinded, end-point (mechanistic, PROBE design).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be masked on their assignment to either the control group vs. registry.
  Assessors for the primary outcome (laboratory measurement) will be blinded to treatment group assigment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eplerenone (Experimental): Patients with MINOCA and an index of microvascular resistance (IMR) greater than or equal to 25 will be randomised to receive eplerenone (starting dose 25 mg, uptitrated to 50mg after two weeks) for six months or standard of care and research protocol study visits. Patients who are screened, give informed consent but are not randomized will enter a followup registry.
  Interventions: Drug: Stratified medicine - Microvascular dysfunction and eplerenone therapy, tablets
- Standard of care (Sham Comparator): Patients with MINOCA and an index of microvascular resistance (IMR) greater than or equal to 25 will be randomised to receive eplerenone (starting dose 25 mg, uptitrated to 50 mg after two weeks) for six months or standard of care and research protocol study visits. Patients who are screened, give informed consent but are not randomized will enter a followup registry.
  Interventions: Other: Stratification and standard care

INTERVENTIONS:
Drug: Stratified medicine - Microvascular dysfunction and eplerenone therapy, tablets — Stratified medicine including interventional diagnostic procedure (IDP) and linked treatment with eplerenone. Patients with an increased IMR (strata with microvascular dysfunction, IMR ≥25) will be eligible for randomization to this arm. Patients randomized to receive eplerenone will be commenced on 25 mg once daily, and uptitrated to 50 mg once daily after two weeks. Treatment will be continued for a period of six months.
  Other Names: Eplerenone
  Arms: Eplerenone
Other: Stratification and standard care — Interventional diagnostic procedure (IDP) without linked treatment i.e., standard care. Patients with an increased IMR (strata with microvascular dysfunction, IMR ≥25) will be eligible for randomization to this arm. In the standard care group, the IDP is performed but the results are not disclosed. The IDP is therefore a sham procedure. Patients randomized to receive eplerenone will be commenced on 25 mg once daily, and uptitrated to 50 mg once daily after two weeks. Treatment will be continued for a period of six months.
  Arms: Standard of care

SUMMARY:
Patients with heart attack or heart injury are tested (angiogram) for blockages in their arteries. Many patients develop heart problems caused by damage to small (microvascular) blood vessels. These issues are also relevant to patients with coronarvirus-19 disease (COVID-19). Eplerenone reduces blood vessel injury and is used to treat heart failure.

Aim: to test the use of eplerenone in patients with heart attack/heart injury who have small vessel disease, including patients with COVID-19

Patients referred to the Golden Jubilee hospital with a suspected heart attack heart / injury will be invited to participate into a registry-based clinical trial. Screening, enrolment and verbal, informed consent will be obtained during the angiogram then written consent on the ward. Small vessel disease will be assessed using a 'diagnostic' guidewire during the standard angiogram. People with small vessel problems will be allocated to a clinical trial of usual care or eplerenone. Coronary microvascular dysfunction is defined as an index of microvascular resistance ≥25. Coronary flow reserve (CFR abnormal <2.0) and resistance reserve ratio (RRR abnormal <2.0), measured simultaneously with IMR, are predefined parameters of interest.

Patients will be allocated into one of the 3 groups:

* Group 1: Patients without coronary microvascular dysfunction. No eplerenone
* Group 2: Patient with coronary microvascular dysfunction. Usual care, no eplerenone.
* Group 3: Small vessels abnormal. Eplerenone tablets.

The primary outcome for the trial will be reduced heart injury (biomarkers) in patients with microvascular disease. We will also test heart function (MRI scan) at enrolment and at six months. All patients (Groups 1, 2 and 3) will have an angiogram. Standard blood tests will be collected during the hospital stay, and then again at 1 and 6 months. Other outcomes include questionnaires (health status). We will gather information on longer-term health outcomes (hospitalisation, death) using confidential electronic record linkage. We will ask for permission to store blood samples for future research.

The research will improve scientific knowledge about eplerenone therapy in this patient group. The study will create a repository of clinical samples and images which will provide vital data for studies of COVID-19.

DETAILED DESCRIPTION:
Background: Myocardial infarction with non-obstructive coronary arteries (MINOCA) involves vascular dysfunction, prognosis is impaired and specific treatments are lacking. Mineralocorticoid antagonist (MRA) therapy attenuates left ventricular remodelling in patients with acute MI without heart failure e.g. REMINDER trial.

Stratified medicine is defined by the Medical Research Council Framework (2015) as the identification of key sub-groups of patients within a heterogeneous population; these being distinguishable groups with differing mechanisms of disease, or particular responses to treatments. Stratification can be used to improve mechanistic understanding of disease processes and enable: the identification of new targets for treatments; the development of biomarkers for disease risk, diagnosis, progression and response to treatment; and treatments to be tested and applied in the most appropriate patient groups.

Objective: To implement stratified medicine in MINOCA.

Hypothesis: In MINOCA, early risk stratification by coronary microvascular dysfunction (index of microvascular resistance (IMR) ≥25) coupled with cardio-protective MRA therapy using eplerenone limits myocardial damage reflected by changes in N-terminal (NT)-pro hormone BNP (NT-proBNP).

Aim: To undertake a developmental clinical study, clarify evidence-gaps and provide training in academic cardiology. Prospective randomized open, blinded end-point (PROBE) design: Step-1: Screening in during coronary angiography of patients with acute myocardial infarction including MINOCA without heart failure or left ventricular ejection fraction ≤40%; Step-2: Guidewire-based measurement of microvascular resistance (culprit artery or if unknown, the left anterior descending coronary artery. Registry population, n=300); Step-3: Stratify subgroup with -increased vascular risk (IMR≥25) (Trial, n=150 eligible for MRA, informed consent); Step-4: Randomise this higher-risk group: eplerenone 25-50 mg daily for 6 months or standard care. Coronary physiology parameters including coronary flow reserve (CFR abnormal <2.0), the resistance reserve ratio (RRR abnormal <2.0) and left ventricular end-diastolic pressure will be prospectively measured.

Outcomes: Primary: within-subject change in NT-proBNP by group; Secondary: left ventricular ejection fraction; left ventricular volumes; patient reported outcome measures (PROMS). Value: Evidence-synthesis on stratified medicine for MINOCA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Acute myocardial infarction or myocardial injury and no obstructive coronary arteries.
* Cardiovascular risk factor (≥1): age >70 years, atrial fibrillation, diabetes, current smoker, eGFR 30 - 60 mL/ minute/1.73 m2, prior MI, treated hypertension or COVID-19 (confirmed or suspected)
* Coronary angiography.

Exclusion Criteria (trial):

* Obstructive coronary artery disease
* Left ventricular ejection fraction ≤40% with evidence of heart failure, following myocardial infarction.
* Estimated glomerular filtration rate <30 mL/ minute/1.73 m2
* Severe liver impairment
* Women who are pregnant, breast-feeding or of child-bearing potential (WoCBP) without a negative pregnancy test and who are unwilling or unable to follow the reproductive restrictions defined in the eligibility criteria and use highly effective contraception as defined in Appendix 2 for the duration of the study treatment and 30 days after last dose of study drug.
* Patients taking one of the following medicines :
* Pre-existing treatment with an MRA :
* Anti-fungal drugs (ketoconazole or itraconazole).
* Antiviral medication (nelfinavir or ritonavir).
* Antibiotics (clarithromycin or telithromycin).
* Nefazodone used to treat depression.
* The combination of an angiotensin converting enzyme (ACE) inhibitor and an angiotensin receptor blocker (ARB)) together.

Exclusion Criteria (registry):

* Contra-indication to cardiovascular magnetic resonance imaging e.g. severe claustrophobia, metallic foreign body.
* Contra-indication to intravenous adenosine, i.e. severe asthma; long QT syndrome; second- or third-degree atrio-ventricular block and sick sinus syndrome.
* Lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Within patient change in NTproBNP | Enrolment, thirty days and six months
  NTproBNP will be measured at enrolment, thirty days and six months

SECONDARY OUTCOMES:
Biomarkers of vascular inflammation | Enrolment, thirty days and six months
  Vascular cell adhesion molecule (VCAM) is a biological marker of vascular inflammation. VCAM will be measured at enrolment, thirty days and six months
Myocardial blood flow at 6 months (MRI) | Performed at six months
  Cardiac MRI with adenosine stress perfusion to measure myocardial blood flow
Health-related quality of life, patient-assessed | Enrolment, thirty days and six months
  European Quality of Life 5-domain 5-Level (EQ-5D-5L) questionnaire, a patient reported outcome measure. Patient assessed score - Scale 0 (worst), 100 (best)
Left ventricular remodelling at 6 months (MRI) | Within fourteen days of enrolment and at six months
  Cardiac MRI performed within fourteen days of enrolment and at six months
Health economics | Enrolment, thirty days and six months
  Institute for Medical Technology Assessment Productivity Cost Questionnaire (iPCQ)
Fibrosis | Enrolment, thirty days and six months
  Circulating (plasma) concentration of procollagen type-I C-terminal pro-peptide (PICP) and collagen type-1 C-terminal telopeptide (CITP) reflect synthesis and degradation of type-I collagen and PICP/CITP ratio reflects collagen turnover.
Haemostasis pathway activation | Enrolment, thirty days and six months
  Circulating (plasma) concentration of factor VIII and other biomarkers of haemostasis pathway activation e.g. D-dimers, fibrinogen

CONTACTS AND LOCATIONS:
Overall Officials: Colin Berry, PhD, Principal Investigator — University of Glasgow
Locations (2):
- United Kingdom (2):
  - University Hospital Hairmyres, East Kilbride, Lanarkshire
  - Golden Jubilee National Hospital, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared based on a bon fide research request and sponsor approval.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: At the end of the study
Access Criteria: Bon fide research request and sponsor approval.

REFERENCES:
- [Background] Collet JP, Thiele H, Barbato E, Barthelemy O, Bauersachs J, Bhatt DL, Dendale P, Dorobantu M, Edvardsen T, Folliguet T, Gale CP, Gilard M, Jobs A, Juni P, Lambrinou E, Lewis BS, Mehilli J, Meliga E, Merkely B, Mueller C, Roffi M, Rutten FH, Sibbing D, Siontis GCM; ESC Scientific Document Group. 2020 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Eur Heart J. 2021 Apr 7;42(14):1289-1367. doi: 10.1093/eurheartj/ehaa575. No abstract available. PMID 32860058
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] Sykes R, Doherty D, Mangion K, Morrow A, Berry C. What an Interventionalist Needs to Know About MI with Non-obstructive Coronary Arteries. Interv Cardiol. 2021 Jun 10;16:e10. doi: 10.15420/icr.2021.10. eCollection 2021 Apr. PMID 34188694
- [Background] Pelliccia F, Pepine CJ, Berry C, Camici PG. The role of a comprehensive two-step diagnostic evaluation to unravel the pathophysiology of MINOCA: A review. Int J Cardiol. 2021 Aug 1;336:1-7. doi: 10.1016/j.ijcard.2021.05.045. Epub 2021 Jun 1. PMID 34087335
- [Background] Ford TJ, Ong P, Sechtem U, Beltrame J, Camici PG, Crea F, Kaski JC, Bairey Merz CN, Pepine CJ, Shimokawa H, Berry C; COVADIS Study Group. Assessment of Vascular Dysfunction in Patients Without Obstructive Coronary Artery Disease: Why, How, and When. JACC Cardiovasc Interv. 2020 Aug 24;13(16):1847-1864. doi: 10.1016/j.jcin.2020.05.052. PMID 32819476
- [Background] Bairey Merz CN, Pepine CJ, Shimokawa H, Berry C. Treatment of coronary microvascular dysfunction. Cardiovasc Res. 2020 Mar 1;116(4):856-870. doi: 10.1093/cvr/cvaa006. PMID 32087007
- [Background] Ford TJ, Stanley B, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, Sidik N, McCartney P, Corcoran D, Collison D, Rush C, McConnachie A, Touyz RM, Oldroyd KG, Berry C. Stratified Medical Therapy Using Invasive Coronary Function Testing in Angina: The CorMicA Trial. J Am Coll Cardiol. 2018 Dec 11;72(23 Pt A):2841-2855. doi: 10.1016/j.jacc.2018.09.006. Epub 2018 Sep 25. PMID 30266608